CLINICAL TRIAL: NCT02940483
Title: Infusion of 5-Azacytidine (5-AZA) Into the Fourth Ventricle or Resection Cavity in Children With Recurrent Posterior Fossa Ependymoma: A Pilot Study
Brief Title: Infusion of 5-Azacytidine (5-AZA) Into the Fourth Ventricle in Children With Recurrent Posterior Fossa Ependymoma
Acronym: 5-AZA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, David Ilan Sandberg, Director of Pediatric Neurosurgery, Professor Pediatric Surgery and Neurosurgery, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0739
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Brain Tumor Recurrent
Keywords: Ependymoma
MeSH Terms: conditions — Brain Neoplasms; Ependymoma | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5-Azacytidine Infusion (Experimental): 12 infusions (once a week) into implanted fourth ventricle catheter/Ommaya reservoir following surgical catheter placement into fourth ventricle.
  Interventions: Drug: 5-Azacytidine

INTERVENTIONS:
Drug: 5-Azacytidine — 5-Azacytidine 10 mg into the fourth ventricle of the brain via the Ommaya reservoir 1 day a week for 12 weeks.
  Other Names: Vidaza, Mylosar

SUMMARY:
The goal of this clinical research study is to establish the safety of direct administration of 5-Azacytidine into the fourth ventricle of the brain or resection cavity in patients with recurrent posterior fossa ependymoma.

DETAILED DESCRIPTION:
If the participant is eligible to take part in this study, the participant will have surgery to place a catheter into the Ommaya reservoir. The Ommaya reservoir is a catheter system that allows drugs to be administered directly to parts of the brain. This catheter will used for the infusion of 5-Azacytidine directly into the 4th ventricle of the brain, which is 1 or the 4 connected fluid-filled cavities in the brain.

If the study doctor thinks it is necessary, based on the location of the tumor, the tumor may also be removed while the participant is already under anesthesia just before the catheter is placed.

Study Drug Administration:

The participant will receive 12 weekly (+/- one day) 10 mg infusions of 5-Azacytidine.

5-Azacytidine will be infused through the Ommaya reservoir catheter directly into the 4th ventricle of the brain starting at a minimum of 7 days after the catheter placement surgery. A MRI will be done to confirm adequate cerebrospinal fluid flow. The 5-Azacytidine infusion will last 2-3 minutes.

If the participant already has an Ommaya catheter, 5-Azacytidine will begin after an MRI has confirmed adequate cerebrospinal fluid flow.

Study Visits:

Prior to first infusion:

Medical history will be reviewed and any updates to health will be recorded. Physical and Neurological exam with vital signs will be done. Blood (about 1 teaspoon) will be drawn for routine test. A lumbar puncture will be done. A MRI scan of the brain and spine will be done to check the status of the disease.

On the days of the 5-Azacytidine Infusion:

A neurological exam with vital signs will be done. A Ommaya reservoir tap (a catheter is placed into the Ommaya reservoir to give the 5-Azacytidine infusion.

Cerebrospinal fluid (about 1 teaspoon) will be collected for routine tests.

Within 7 days of completing the Final infusion:

A neurological exam with vital signs will be done. A lumbar puncture will be done. A MRI scan of the brain and spine will be done to check status of the disease.

Length of Study:

The participant will receive 12 infusions of 5-Azacytidine, as long as the doctor thinks it is in their best interest. The participant will no longer be able to receive the study drug if the disease gets worse, if intolerable side effects occur, or if unable to follow study directions.

This is an investigation study. 5-Azacytidine is FDA approved and commercially available to be given subcutaneous or into the bloodstream (intravenously) but has never been given in the 4th ventricle of the brain. The infusion of 5-Azacytidine into the 4th ventricle of the brain is investigational.

Up to 10 patients will be enrolled in this study. All will be enrolled at Children's Memorial Hermann Hospital

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Patients with histologically verified ependymoma, with recurrence or progression involving anywhere in the brain and/or spine. To be eligible, patients' disease must have originated in the posterior fossa of the brain.
* Patient must have either measurable or evaluable tumor as assessed by MRI of the brain and total spine.
* An implanted catheter in the fourth ventricle or posterior fossa tumor cavity attached to a ventricular access device or agreement to have one placed.
* A minimum of 7 days between last dose of systemic chemotherapy and/or radiation therapy and first infusion of 5-Azacytidine into fourth ventricle.
* Life expectancy of at least 12 weeks in the opinion of the PI
* Lansky score of 50 or greater if ≤16 years of age or Karnofsky score of 50 or greater if > 16 years of age.
* Existing neurological deficits must have been stable for a minimum of 1 week prior to study enrollment.
* Patients must have recovered from the acute toxic effects of all prior anticancer chemotherapy
* Adequate bone marrow function defined by peripheral absolute neutrophil count (ANC) ≥ 500/µL, platelet count ≥ 50,000/ µL (transfusion independent), and hemoglobin ≥9.0 gm/dL (may receive RBC transfusions)
* Patient or patient's legal representative, parent(s), or guardian able to provide written informed consent.

Exclusion Criteria:

* Enrolled in another treatment protocol
* Has received another investigational or chemotherapy agent or radiation therapy within 7 days prior to 5-Azacytidine infusion into the fourth ventricle.
* Evidence of untreated infection
* Pregnant of lactating women

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with grade 3 through grade 5 new neurological adverse events that are related to study drug, graded according to NCI CTCAE Version 4.0 | 4 months
  New neurological deficit defined as new cranial neuropathy, nystagmus, change in mental status, motor deficit or cerebellar finding (ataxia, dysmetria, dysdiadochokinesis) that is attributed by treating physicians to intraventricular 5-Azacytidine infusions. Primary endpoint for basis of safety monitoring is acute toxicity occurring at any time within 30 days of receiving the intraventricular 5-Azacytidine infusion. Rate of acute toxicity monitored using Bayesian method of Thall and Sung. Method of Kaplan and Meier used to estimate unadjusted distributions o time to a neurological deficit and progression free survival time and summary statistic of all variable computed and tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: David I Sandberg, M.D., Principal Investigator — UTHealth
Locations (1):
- UTHealth & Children's Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lang F, Liu Y, Chou FJ, Yang C. Genotoxic therapy and resistance mechanism in gliomas. Pharmacol Ther. 2021 Dec;228:107922. doi: 10.1016/j.pharmthera.2021.107922. Epub 2021 Jun 23. PMID 34171339